CLINICAL TRIAL: NCT00000869
Title: A Phase III Randomized, Blinded Study of Nevirapine for the Prevention of Maternal-Fetal Transmission in Pregnant HIV-Infected Women
Brief Title: A Study of Nevirapine for the Prevention of HIV Transmission From Mothers to Their Babies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 316; 11290 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy Trimester, Third; Placebos; Pregnancy; Pregnancy Complications, Infectious; Administration, Oral; Nevirapine; Disease Transmission, Vertical; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious | interventions — Nevirapine

INTERVENTIONS:
Drug: Nevirapine

SUMMARY:
The purpose of this study is to see if giving the anti-HIV drug nevirapine (NVP) to HIV-positive pregnant women and their babies can help reduce the chance that a mother will give HIV to her baby during delivery. This study will also test the safety of the drug and see how well it is tolerated by the mother and her baby.

Previous studies suggest that NVP is a promising medication for blocking HIV transmission from HIV-positive mothers to their babies.

DETAILED DESCRIPTION:
Nevirapine has several properties that make it an attractive candidate for antiretroviral therapy to interrupt HIV-1 transmission in the intrapartum and early postpartum period. The pharmacokinetic profile suggested that nevirapine would be rapidly absorbed and transferred to the infant in utero when given during labor and delivery. In addition, nevirapine has been shown to penetrate cell-free virions and inactivate virion-associated reverse transcriptase (RT) in situ. This property would be potentially useful in inactivating cell-free virions in the genital tract as well as in breast milk. These characteristics of nevirapine suggest that treatment of an HIV-infected pregnant woman in labor with an oral dose of nevirapine may provide a prophylactic level of nevirapine in the infant during the time of exposure to virus in the birth canal and/or maternal blood. In addition, nevirapine may inactivate the virion-associated RT present in cell-free virions in the genital tract or breast milk.

Women are randomized to receive either NVP or the corresponding placebo in active labor. Women are randomized at any time after their 32nd week gestation [AS PER AMENDMENT 1/13/98: 28th week gestation] [AS PER AMENDMENT 2/23/00: 20th week gestation]. The randomization is stratified using two factors: (1) use of [AS PER AMENDMENT 2/23/00: current or anticipated] antiretroviral therapy during the current pregnancy (no therapy at all; monotherapy for any duration; multi-agent therapy for any duration), and (2) CD4 cell count at the time of randomization (less than 200 cells; 200 - 399 cells; 400 cells or greater). Mothers are followed on study for 4 to 6 weeks postpartum. Mothers are also encouraged to follow the regimen of zidovudine (ZDV) outlined in the Office of Public Health and Science (PHS) treatment guidelines for both themselves and their infants. Infants are administered either NVP or placebo between 48 and 72 hours of life. The infant's study drug is the same as the mother's randomized treatment assignment. Infants are dosed with the study drug according to their randomization group regardless of whether the mother received the study drug. Infants are followed for 4 to 6 weeks, and are tested for HIV at 4 to 6 weeks, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria

Women may be eligible for this study if they:

* Are HIV-positive.
* Are at least 20 weeks pregnant. (This study has been changed. Women no longer have to be 28 weeks pregnant.)
* Have consent from the child's father (if available).
* Are at least 13 years old (consent of parent or guardian required if under 18).

Exclusion Criteria

Women will not be eligible for this study if they:

* Have ever taken NNRTIs (nonnucleoside reverse transcriptase inhibitors).
* Are enrolled in another pregnancy treatment study.
* Are allergic to benzodiazepines.
* Have liver disease.
* Plan to breast-feed.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2009
Dates: Study Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Dorenbaum, Study Chair; John Sullivan, Study Chair
Locations (72):
- United States (69):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - Univ of South Alabama, Mobile, Alabama
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - San Francisco Gen Hosp, San Francisco, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Children's Hosp of Denver, Denver, Colorado
  - Connecticut Children's Med Ctr, Farmington, Connecticut
  - Univ of Connecticut / Farmington, Farmington, Connecticut
  - Washington Hosp Ctr, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Univ of Florida Gainesville, Gainesville, Florida
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami / Jackson Memorial Hosp, Miami, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Med College of Georgia, Augusta, Georgia
  - The Med Ctr Inc, Columbus, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Tulane Univ Hosp of New Orleans, New Orleans, Louisiana
  - Univ Hosp, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - Cooper Hosp - Univ Med Ctr / UMDNJ - New Jersey Med Schl, Camden, New Jersey
  - UMDNJ - Robert Wood Johnson Med School / Pediatrics, New Brunswick, New Jersey
  - St Peter's Med Ctr, New Brunswick, New Jersey
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Saint Joseph's Hosp and Med Ctr/UMDNJ - New Jersey Med Schl, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Metropolitan Hosp Ctr, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of North Carolina at Chapel Hill / Duke Univ Med Ctr, Durham, North Carolina
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Hosp of the Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Temple Univ School of Medicine, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Regional Med Ctr at Memphis, Memphis, Tennessee
  - Methodist Hosp Central, Memphis, Tennessee
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Children's Hosp of the King's Daughters, Norfolk, Virginia
  - Senetara Norfolk Gen Hosp, Norfolk, Virginia
  - Med College of Virginia, Richmond, Virginia
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
  - Tacoma Gen Hosp, Tacoma, Washington
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] Cunningham CK, Britto P, Gelber R, Dorenbaum A, Mofenson L, Culnane M, Sullivan JL. Genotypic resistance analysis in women participating in PACTG 316 with HIV-1 RNA >400 copies/ml. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 712)
- [Background] Mirochnick M, Dorenbaum A, Cunningham-Schrader B, Cunningham C, Gelber R, Mofenson L, Sullivan J. Cord blood protease inhibitor (PI) concentrations in infants born to mothers receiving PIs. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 710)
- [Background] Dorenbaum A. Report of results of PACTG 316: an international phase III trial of standard antiretroviral (ARV) prophylaxis plus nevirapine (NVP) for prevention of perinatal HIV transmission. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no LB7)
- [Background] Cunningham CK, Chaix ML, Rekacewicz C, Britto P, Rouzioux C, Gelber RD, Dorenbaum A, Delfraissy JF, Bazin B, Mofenson L, Sullivan JL. Development of resistance mutations in women receiving standard antiretroviral therapy who received intrapartum nevirapine to prevent perinatal human immunodeficiency virus type 1 transmission: a substudy of pediatric AIDS clinical trials group protocol 316. J Infect Dis. 2002 Jul 15;186(2):181-8. doi: 10.1086/341300. Epub 2002 Jun 26. PMID 12134253
- [Background] Mirochnick M, Dorenbaum A, Blanchard S, Cunningham CK, Gelber RD, Mofenson L, Culnane M, Sullivan JL. Predose infant nevirapine concentration with the two-dose intrapartum neonatal nevirapine regimen: association with timing of maternal intrapartum nevirapine dose. J Acquir Immune Defic Syndr. 2003 Jun 1;33(2):153-6. doi: 10.1097/00126334-200306010-00006. PMID 12794547
- [Background] Cunningham CK, Balasubramanian R, Delke I, Maupin R, Mofenson L, Dorenbaum A, Sullivan JL, Gonzalez-Garcia A, Thorpe E, Rathore M, Gelber RD. The impact of race/ethnicity on mother-to-child HIV transmission in the United States in Pediatric AIDS Clinical Trials Group Protocol 316. J Acquir Immune Defic Syndr. 2004 Jul 1;36(3):800-7. doi: 10.1097/00126334-200407010-00006. PMID 15213563
- [Background] Watts DH, Balasubramanian R, Maupin RT Jr, Delke I, Dorenbaum A, Fiore S, Newell ML, Delfraissy JF, Gelber RD, Mofenson LM, Culnane M, Cunningham CK; PACTG 316 Study Team. Maternal toxicity and pregnancy complications in human immunodeficiency virus-infected women receiving antiretroviral therapy: PACTG 316. Am J Obstet Gynecol. 2004 Feb;190(2):506-16. doi: 10.1016/j.ajog.2003.07.018. PMID 14981398
- [Result] Newell ML, Huang S, Fiore S, Thorne C, Mandelbrot L, Sullivan JL, Maupin R, Delke I, Watts DH, Gelber RD, Cunningham CK; PACTG 316 Study Team. Characteristics and management of HIV-1-infected pregnant women enrolled in a randomised trial: differences between Europe and the USA. BMC Infect Dis. 2007 Jun 20;7:60. doi: 10.1186/1471-2334-7-60. PMID 17584491